CLINICAL TRIAL: NCT00636233
Title: The Hereditary Basis of Neural Tube Defects
Brief Title: Genetics of Spina Bifida and Anencephaly
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00016517; R01NS039818 (NIH)
Record Dates: First submitted 2008-03-09; First posted 2008-03-14 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2019-03

CONDITIONS: Anencephaly; Acrania
Keywords: anencephaly; acrania
MeSH Terms: conditions — Anencephaly; Neural Tube Defects

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, saliva, cord blood, fetal tissue, cultured fetal cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anencephaly: Fetuses with anencephaly, parents and siblings

SUMMARY:
The goal of this research study is to discover the genetic and environmental factors that contribute to the cause of neural tube defects such as spina bifida and anencephaly. Ultimately, this type of research may result in improved diagnosis, improved treatment and possibly prevention.

ELIGIBILITY:
Not currently enrolling new participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any current pregnancy affected by anencephaly or acrania.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1993-05; Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
genetic factors associated with neural tube defects | end of the study
  This study aims to discover genetic factors associated with neural tube defects such as anencephaly.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Ashley-Koch, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Anencephaly study description — http://dmpi.duke.edu/anencephaly
- See also: Neural tube defect study description — http://dmpi.duke.edu/neural-tube-defects-ntds